CLINICAL TRIAL: NCT02492412
Title: Multi-center, Randomized, Double-blind, Active Comparator- Controlled, Parallel Study Evaluating the Efficacy and Safety of HE10 in Subjects With Dry Eye Syndrome
Brief Title: Efficacy and Safety of HE10 for Dry Eye Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Huons
Record Dates: First submitted 2015-06-25; First posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins; Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HE10 (Experimental): Drug: HE10 1~2 drops b.i.d at 12 hour interval for 12 weeks
  Interventions: Drug: HE 10
- Restasis (Active Comparator): Drug: Restasis(Cyclosporine 0.05%) 1~2 drops b.i.d at 12 hour interval for 12 weeks
  Interventions: Drug: Restasis

INTERVENTIONS:
Drug: HE 10
  Arms: HE10
Drug: Restasis
  Other Names: 0.05% cyclosporine
  Arms: Restasis

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of HE10 eye drop for the patients with moderate to severe dry eye syndrome.

DETAILED DESCRIPTION:
This study is to compare the efficacy and safety of HE10 and Restasis for patients with moderate to severe dry eye syndrome in multi-center, double-blind, randomized, active comparator-controlled, parallel design, non-inferiority Phase III clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Corneal staining score of ≥2(Oxford grade)
* Schirmer test score (without anesthesia) < 10 mm/5 min in either eye
* Tear break-up time is 10 seconds or less
* Screening both eyes, the corrected visual acuity is 0.2 or more

Exclusion Criteria:

* Current or recent patients used dry eye syndrome medications (topical or systemic) that may affect the status
* The patients with systemic or ocular disorders affected the test result
* Being treated with systemic steroid
* History of eyeball surgical operation within 3 months of screening visit
* Wearing contact lenses within 2 weeks of screening visit
* Be a use or used punctual plug within 1 month of screening vist
* Use of cyclosporine eye drop within 3 weeks
* Pregnancy or Breastfeeding
* Intraocular pressure > 25 mmHg
* Abnormal eyelid function : Disorders of the eyelids or eyelashes

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Corneal staining Test to assess eye dryness | 12 weeks
  Change from baseline in eye dryness at 12 weeks